CLINICAL TRIAL: NCT07335536
Title: The Efficacy of Remimazolam on Incidence of Hypoxia During Sedated Transvaginal Oocyte Retrieval: A Multicenter Randomized Controlled Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diansan Su (Other)
Responsible Party: Sponsor-Investigator, Diansan Su, Director of Anesthesiology, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJU2025C086
Record Dates: First submitted 2025-09-22; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hypoxia; Infertility; Infertility Assisted Reproductive Technology
Keywords: Hypoxia; oocyte retrieval; remimazolam; general anesthesia
MeSH Terms: conditions — Hypoxia; Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol-alfentanil (Active Comparator): Sedation using remimazolam-alfentanil
  Interventions: Drug: propofol-alfentanil
- remimazolam-alfentanil (Experimental): Sedation using remimazolam-alfentanil
  Interventions: Drug: remimazolam-alfentanil combination

INTERVENTIONS:
Drug: remimazolam-alfentanil combination — Administer 7 μg/kg of fentanyl first，then given remimazolam 0.2 mg/kg (1-minute bolus), followed by 1 mg/kg/h infusion.
  Arms: remimazolam-alfentanil
Drug: propofol-alfentanil — Administer 7 μg/kg of fentanyl first，then given propofol 2 mg/kg (1-minute bolus), followed by 6 mg/kg/h infusion.
  Arms: propofol-alfentanil

SUMMARY:
Hypoxia is the most common adverse reaction during sedation outside the operating room.Exploring novel drug combinations to reduce the incidence of hypoxia during sedation in patients undergoing transvaginal oocyte retrieval procedures enhances patient safety and lowers perioperative adverse event rates. This multicenter, prospective, randomized, controlled clinical study will compare the hypoxia incidence rate of the remimazolam-alfentanil combination against the commonly used propofol-alfentanil combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 50 years planning to undergo painless oocyte retrieval
* Subjects classified as American Society of Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* Subjects with contraindications to general anesthesia, acute or severe cardiovascular disease history, acute upper respiratory infection, chronic obstructive pulmonary disease (COPD), asthma attacks, or uncontrolled hypertension
* Subjects with alcohol abuse
* Subjects with severe hepatic or renal insufficiency, severe cardiovascular disease, or psychiatric disorder history
* Subjects with hearing impairment preventing communication
* Subjects with a history of long-term sedative or opioid use, or allergies to benzodiazepines, flumazenil, opioids and their antidotes, propofol, eggs, or soy products
* Subjects with SpO2 < 95% while breathing room air after entering the room

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO₂ between 75% and 89% with duration <60 seconds

SECONDARY OUTCOMES:
Incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s
Incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO₂ < 95%
Proportion of hypoxic correction measures | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Corrective measures for hypoxia should be implemented in the following sequence: increase oxygen flow rate, perform jaw thrust, administer positive pressure ventilation via a face mask, insert a nasopharyngeal airway while performing jaw thrust, and proceed to endotracheal intubation or mechanical ventilation with a laryngeal mask until SpO₂ reaches ≥95%.

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang F, Chang H, Qing W, Yu R, Liao Q, Tong J. Remimazolam Tosylate Combined with Low-Dose Propofol Improves Sedation and Safety in Hysteroscopy. Drug Des Devel Ther. 2022 Nov 29;16:4101-4108. doi: 10.2147/DDDT.S390403. eCollection 2022. PMID 36471692